CLINICAL TRIAL: NCT05486507
Title: The Health Benefits of Montmorency Tart Cherry Juice Supplementation in Adults With Mild to Moderate Ulcerative Colitis; a Placebo Randomized Control Trial
Brief Title: Health Benefits of Tart Cherry in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tart cherry ulcerative colitis
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montmorency tart cherry juice (Experimental)
  Interventions: Dietary Supplement: Montmorency tart cherry
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Montmorency tart cherry — US grown Montmorency tart cherry 60ml per day for 6 weeks.
  Arms: Montmorency tart cherry juice
Dietary Supplement: Placebo — Taste matched placebo.
  Arms: Placebo

SUMMARY:
Ulcerative Colitis (UC) is a long-term inflammatory condition of the digestive tract. People with UC often have unpredictable and debilitating symptoms, including abdominal pain, diarrhoea and fatigue. In addition, they require long-term treatment with frequent negative effects, the need of surgery and hospitalisations. Therefore, people with UC report a lower health-related quality of life (HRQOL) compared with healthy individuals. The most common medication for inflammatory bowel disease is a strong immunosuppressant which has previously (in 2017) been found to be the most expensive medication prescribed at hospitals in the NHS. Unfortunately, biologics has a lot of negative side effects and thus reducing the need of them in patients can benefit both the NHS as a whole by reducing the cost and improving the quality of life of patients by reducing the unwanted side effects of the biologics. Supplementation of Montmorency tart cherry juice might be a simple, safe, and low-cost intervention for improving symptoms in patients with UC. This is because it has the potential to naturally reduce inflammation in the digestive system and thus improve symptoms. Research in animal models has shown a potential for improvement in physiological responses with similar supplements including blueberries, black raspberries and even Montmorency tart cherries, with only one study in human participants exploring bilberry supplementation.

However, despite anthocyanins concentrations from Montmorency tart cherries being superior to other berries, dietary interventions using tart cherry supplementation for UC have not received any attention in human participants. The primary purpose of the proposed investigation is to undertake a placebo randomized control trial examining the ability of a Montmorency tart cherry juice supplement to provide symptom relief and health related wellbeing outcomes in those with mild to moderately active UC and to understand the biological mechanisms behind any changes in symptoms.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of UC for at least 6 months
* Current mild to moderate disease activity
* Age between 18 and 65 years
* Stable use of medication for at least 3 months respectively.

Exclusion Criteria:

* Diabetes
* HIV
* Hepatitis B and C infection
* Abscesses
* Unstable medical conditions that would likely prevent the subject from completing the study
* Food allergies to cherries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Quality of Life Questionnaire | This parameter will be examined at baseline.
  The scale has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health).
Inflammatory Bowel Disease Quality of Life Questionnaire | This parameter will be examined at 6 weeks.
  The scale has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health).

SECONDARY OUTCOMES:
Simple clinical colitis activity index | This parameter will be examined at baseline.
  The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
Simple clinical colitis activity index | This parameter will be examined at 6 weeks.
  The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
Hospital anxiety and depression scale | This parameter will be examined at baseline.
  The Hospital Anxiety and Depression Scale measures anxiety and depression in patients. A higher score indicates greater anxiety and depression.
Hospital anxiety and depression scale | This parameter will be examined at 6 weeks.
  The Hospital Anxiety and Depression Scale measures anxiety and depression in patients. A higher score indicates greater anxiety and depression.
European Quality of Life Scale | This parameter will be examined at baseline.
  The European Quality of Life Scale is an instrument for measuring quality of life across patient groups and cultures and is conceptually distinct from health status or other causal indicators of quality of life. A higher score indicates higher quality of life.
European Quality of Life Scale | This parameter will be examined at 6 weeks.
  The European Quality of Life Scale is an instrument for measuring quality of life across patient groups and cultures and is conceptually distinct from health status or other causal indicators of quality of life. A higher score indicates higher quality of life.
International Physical Activity Questionnaire - Short Form | This parameter will be examined at baseline.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) addresses the number of days and time spent on physical activity in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days. The IPAQ-SF sum score is expressed in physical activity Metabolic Equivalent of Task minutes per day or week.
International Physical Activity Questionnaire - Short Form | This parameter will be examined at 6 weeks.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) addresses the number of days and time spent on physical activity in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days. The IPAQ-SF sum score is expressed in physical activity Metabolic Equivalent of Task minutes per day or week.
IBD Fatigue Scale | This parameter will be examined at baseline
  The IBD Fatigue Scale is comprised of two components. Part 1 the questionnaire will identify fatigue, its severity, frequency and duration and scores range from 0-20 with a higher score meaning greater fatigue. Part 2 assesses the perceived impact of fatigue on your daily activities and scores range from 0-120 with a higher score meaning greater perceived impact.
IBD Fatigue Scale | This parameter will be examined at 6 weeks
  The IBD Fatigue Scale is comprised of two components. Part 1 the questionnaire will identify fatigue, its severity, frequency and duration and scores range from 0-20 with a higher score meaning greater fatigue. Part 2 assesses the perceived impact of fatigue on your daily activities and scores range from 0-120 with a higher score meaning greater perceived impact.
Gut bacteria and fungi Gut bacteria and fungi | This parameter will be examined at baseline
  Gut bacteria and fungi will be measured from feacal samples with higher values indicating greater levels of bacteria and fungi in the gut.
Gut bacteria and fungi | This parameter will be examined at 6 weeks.
  Gut bacteria and fungi will be measured from feacal samples with higher values indicating greater levels of bacteria and fungi in the gut.
TNF alpha | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
TNF alpha | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-6 | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-6 | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-17A | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-17A | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-12 | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-12 | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-23 | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-23 | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-10 | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Interleukin-10 | This parameter will be examined at 6 weeks.
  This measure will be obtained from blood samples to provide a measure of inflammation.
Transforming growth factor Beta | This parameter will be examined at baseline
  This measure will be obtained from blood samples to provide a measure of inflammation.
Transforming growth factor Beta | This parameter will be examined at 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Central Lancashire, Preston, Lancashire
  - University of Hertfordshire, London